CLINICAL TRIAL: NCT00926354
Title: Phase II Open Study to Evaluate Safety and Efficacy of AS101 for the Treatment of Thrombocytopenia in Solid Tumor
Brief Title: Application of AS101 for the Treatment of Thrombocytopenia in Solid Tumor Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's considerations
Sponsor: BioMAS Ltd (Industry)
Responsible Party: BioMas LTD, BioMas LTD
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #71 REV 00
Record Dates: First submitted 2009-06-17; First posted 2009-06-23 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2011-06

CONDITIONS: Chemotherapy Induced Thrombocytopenia
MeSH Terms: interventions — ammonium trichloro(dioxoethylene-O,O'-)tellurate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AS101 infusion (Experimental): Twenty patients who developed thrombocytopenia after a chemotherapy course will receive i.v. infusions of 3mg/m2 AS101 twice a week in addition to the standard chemotherapy regimen, during the following 4 chemotherapy courses.
  Interventions: Drug: AS101
- Control group (No Intervention): Twenty patients who developed thrombocytopenia during chemotherapy course will be treated according to standard of care and will not receive the investigational product. Their medical condition will be followed and a complete blood count will be performed routinely once weekly.

INTERVENTIONS:
Drug: AS101 — intravenous infusions of 3mg/m2 AS101 twice a week in addition to the standard chemotherapy regimen during the following 4 chemotherapy courses.
  Arms: AS101 infusion

SUMMARY:
Chemotherapy Induced Thrombocytopenia is a common side-effect of bone marrow suppression as a result of a chemotherapy treatment. AS101 is a tellurium based small compound with immunomodulating characteristics which attributed to the direct inhibition of the anti-inflammatory cytokine IL-10. AS101 was previously shown to induce a significant reduction in thrombocytopenia that accompany cancer therapy with no major toxicity . This phase II randomized open study will evaluate the efficacy of AS101 for the treatment of chemotherapy induced thrombocytopenia in patients with various solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Appropriate histology of solid tumors.
* Platelet counts < 70,000/μl.
* Performance Status (PS) of 0-2
* Adequate renal function: Serum creatinine ≤1.5 mg/dL
* Adequate liver function: Serum (total) bilirubin ≤ 1.5 ULN. AST, ALT ≤ 2.5 x ULN in patients without liver metastases, ≤ 5 x ULN in patients with liver metastases. Albumin ≥ 2.5 g/dL (Only for patients who will receive AS101).
* INR ≤ 1.5 and PTT ≤ 1.5 x ULN (Only for patients who will receive AS101).

Exclusion Criteria:

* Patients unable to provide fully informed consent.
* Women who are pregnant or breast feeding.
* The patient is participating in another trial of an investigational drug or has done so within 28 days prior to the pre-treatment visit.
* The patient has congestive heart failure-New York Heart Association (CHF-NYHA) grade II or higher, and/or myocardial infarction within the last 12 months, or any cardiac disorder which in the opinion of the Investigator would put the patient at risk.
* The patient has a history of chronic alcohol or drug abuse within the last 5 years.
* The patient has any other clinically significant medical condition, psychiatric condition or laboratory abnormality which would, in the judgment of the Investigator, interfere with the patient's ability to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Incidence of thrombocytopenia events (platelets <70,000) over the study period of the study groups | continously during study and 6 months after study termination

SECONDARY OUTCOMES:
Evaluation of Safety and tolerability; Thrombocytopenia events that caused treatment delays and chemotherapy dose; reductions; Progression Free Survival (PFS); Response Rate (RR); | continously during study and 6 months after study termination

CONTACTS AND LOCATIONS:
Overall Officials: Baruch Klein, Prof, Principal Investigator — Meir Medical Center, Kfar Saba, Israel
Locations (1):
- Meir Medical Center, Kfar Saba, Israel